CLINICAL TRIAL: NCT00676572
Title: p38 MAPK Activation as the Basis for Corticosteroid Insensitivity in Severe Asthma
Brief Title: p38 Mitogen-Activated Protein Kinase (MAPK) and Steroid Insensitivity in Asthma
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Fan Chung, Professor, Imperial College London
Other Study IDs: 08/H0708/29; CRO1014
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Asthma
Keywords: severe asthma; corticosteroid insensitivity
MeSH Terms: conditions — Asthma | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sputum cell pellets and supernatant; BAL supernatant; endobronchial biopsies; smooth muscle cell culture from biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe asthma
  Interventions: Other: Fiberoptic bronchoscopy; blood test
- Non-severe asthma
  Interventions: Other: Fiberoptic bronchoscopy; blood test

INTERVENTIONS:
Other: Fiberoptic bronchoscopy; blood test — Fiberoptic bronchoscopy for obtention of alveolar macrophages and bronchial biopsies for histology and culture of airway smooth muscle cells

SUMMARY:
This research aims to find out how the inflammation in patients suffering from severe asthma is different from that in non-severe asthma, and how it may prevent corticosteroids from working efficiently in severe asthma.

It will look,in particular, at a protein enzyme called p38 mitogen-activated protein kinase (p38 MAPK for short)which controls the activation of several important pathways in the cell. We wish to find out whether this enzyme is more active in cells obtained from patients with severe asthma compared to those with non-severe asthma. We would like to understand how this enzyme can cause the cell to respond less well to the anti-inflammatory effects of corticosteroids. We also wish to find out whether any specific inhibitors of p38 MAPK can improve severe asthma by improving the effects of corticosteroids on these cells.

We hypothesise that activation of the intracellular MAPK signalling pathway underlies the inflammatory processes of severe asthma, and leads to the diminution of the anti-inflammatory actions of CS through histone modification.

DETAILED DESCRIPTION:
DESIGN Comparative study to analyse differences in the characteristics of lung macrophages and blood monocytes between non-severe and severe asthmatics.

AIMS

1. To determine whether there are differences in terms of cell expression and activation between lung macrophages and blood monocytes from non-severe and severe asthma
2. To determine the mechanisms of the lung macrophage and blood monocyte relative resistance to the effect of corticosteroids in severe asthma, and particularly focus on the role of p38 MAPK
3. To determine the differences in airway smooth muscle cells between non-severe and severe asthma

OUTCOME MEASURES

1. Clinically the differences in inflammatory and remodelling markers between non-severe and severe asthma
2. Differences in histone phosphorylation, NF-kB activity and glucocorticoid receptor activation and actions in macrophages and monocytes between non- severe and severe asthma
3. Differences in behaviour of airway smooth muscle cells cultured from biopsies obtained from non-severe and severe asthma

Severe and non-severe asthmatic subjects will be classified following ATS criteria. They undergo spirometry with reversibility testing, PC20, skin prick tests, exhaled nitric oxide measurements and induced sputum. They will have blood taken for PBMCs and undergo fiberoptic bronchoscopy for obtention of alveolar macrophages and bronchial biopsies

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Physician diagnosis of asthma

Non-severe asthmatic subjects:

* mild to moderately severe asthma.
* The groups will be defined as follows, according to their need for treatments (as established in the Asthma Management GINA or BTS guidelines):

  1. Mild: intermittent symptoms and need for reliever bronchodilator less than once a day
  2. moderate asthma: well-controlled asthma with minimal symptoms while on inhaled corticosteroid therapy not exceeding 2,000 μg beclomethasone equivalent.

Severe asthmatic subjects:

* will have at least 1 major and 2 minor criteria (as below) Major characteristics (at least one of the following criteria)

  * Treatment with continuous or near continuous (>50% of year) oral corticosteroids
  * Requirement for treatment with high dose inhaled corticosteroids (ICS) Minor characteristics (at least 2 out of the following)

    1. Requirement for daily treatment with a controller medication in addition to ICS e.g. LABA, theophylline, leukotriene antagonist
    2. Asthma symptoms requiring SABA on a daily or near daily basis
    3. Persistent airways obstruction (FEV1 <80% predicted, diurnal PEF variation >20%)
    4. One or more emergency care visits for asthma per year
    5. 3 or more steroid "bursts" per year
    6. Prompt deterioration with ≤ 25% reduction in oral or ICS
    7. Near fatal asthma event in the past

Exclusion Criteria:

* Current smokers, or less than 3 years since quitting smoking (< 5 pack/years)
* Less than 4 weeks from an exacerbation
* On steroid-sparing agent or immunosuppressant such as azathioprine, methotrexate and ciclosporin
* Concomitant anti-IgE therapy
* On anti-platelet or anti-coagulant drugs
* Low platelet count
* Pregnancy or breast-feeding
* Intubation for asthma within 6 months of entry into this study (if undergoing bronchoscopy)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Asthmatic subjects will be recruited from asthma clinics at the Royal Brompton Hospital and from primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian F Chung, MBBS MD FRCP DSc, Principal Investigator — Imperial College London; Pankaj Bhavsar, BSc PhD, Principal Investigator — Imperial College London
Locations (1):
- Asthma Laboratory, Royal Brompton Hospital, Sydney Street, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bhavsar P, Khorasani N, Hew M, Johnson M, Chung KF. Effect of p38 MAPK inhibition on corticosteroid suppression of cytokine release in severe asthma. Eur Respir J. 2010 Apr;35(4):750-6. doi: 10.1183/09031936.00071309. Epub 2009 Oct 19. PMID 19840967

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Severe Asthma | Non-severe Asthma
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Asthma | Non-severe Asthma | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (2.67) | 32.8 (3.88) | 39.9 (3.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 1 | 3 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Differences in Activity and Downstream Activity of the p38 MAPK Activity in Macrophages or PBMCs Between Those From Severe and Non-Severe Asthmatics
Time Frame: 3 years
Population: Data no collected
Arm/Group | Severe Asthma | Non-severe Asthma
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Differences in the Effect of p38 MAPK Inhibitor in Dexamethasone-Inhibition of Cytokine Release From Alveolar Macrophages and PBMCs Between Severe and Non-Severe Asthmatics
Description: Percentage of Suppression of IL6 release by p38 MAPK inhibitor
Time Frame: 3 years
Measure: Mean (Standard Error); unit: percentage of suppression of IL6 release
Arm/Group | Severe Asthma | Non-severe Asthma
Number analyzed (Participants) | 6 | 6
percentage of suppression of IL6 release | 50 (20) | 8 (10)
Statistical Analysis 1: Comparison: Severe Asthma vs Non-severe Asthma; Test type: Superiority; p < 0.05, t-test, 2 sided — calculated p values

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Severe Asthma | Non-severe Asthma
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes